CLINICAL TRIAL: NCT00457236
Title: Impact of the Degree of Peri-Interventional Platelet Inhibition After Loading With Clopidogrel on Early Clinical Outcome of Elective Coronary Stent Placement
Brief Title: Effect of Clopidogrel Loading and Risk of PCI
Acronym: EXCELSIOR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Other Study IDs: HZ-BK-2003-1
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Artery Disease; Drug Resistance
Keywords: Clopidogrel; Coronary Artery Disease; Dose-Response Relationship, Drug; Drug Resistance; PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This study is a prospective, single-center evaluation of the impact of the variability in platelet response after loading with clopidogrel on the peri-interventional risk of patients undergoing PCI.

DETAILED DESCRIPTION:
Background: Platelet responses after loading with clopidogrel are highly variable. The impact of this variability on the peri-interventional risk of patients undergoing PCI has not been investigated prospectively.

Objectives: Our prospective study test the hypothesis that the 30-day clinical outcome of elective percutaneous catheter intervention (PCI) differs between strata defined by quartiles of platelet aggregation after loading with 600mg of clopidogrel. Further on we will investigate impact of the variability in platelet response on long-term outcome after PCI.

Methods: Our study will include consecutive patients undergoing elective coronary stent placement. Before PCI, patients receive a loading dose of 600mg of clopidogrel followed by 75mg daily. Primary end point is the 30-day composite of death, myocardial infarction and target lesion revascularization (MACE). Platelet aggregation was assessed immediately before PCI by optical aggregometry (5µmol/L ADP).

Sample size calculation was based on ISAR-REACT which comprised a cohort with similar selection criteria and treatment strategy. Thus, we assume an incidence of the primary end point of 4.2%. We design our study to test the hypothesis that the incidence of the primary end point differed by quartiles of ADP-induced platelet aggregation. We intend to have a power of 0.80 to detect an effect size of 0.015 (for example 3-fold risk in 4th quartile) with a 2-sided P-value less than 0.05. With these assumptions we obtain a sample size of at least 748 and aime for a cohort of 800.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary stenting
* Pretreatment with a bolus dose of 600mg of clopidogrel prior to coronary stent implantation
* Pretreatment with aspirin ≥ 100 mg per day for at least 7 days
* Age > 18 years
* Written consent

Exclusion Criteria:

* Troponin T on admission > 0.03 ng/mL
* Myocardial infarction or fibrinolytic therapy within the previous 14 days
* Cardiogenic shock
* Contraindication for aspirin or clopidogrel
* Oral anticoagulation
* Pretreatment with heparin or a thienopyridine within the previous 14 days
* Use of a GP IIb/IIIa-receptor antagonist during PCI
* Platelet count < 100.000/µl
* Severe disorders of the coagulation system
* Severe impairment of liver or kidney function
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2003-03; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Franz-Josef Neumann, MD, Study Director — Heart Center Bad Krozingen, Germany
Locations (1):
- Heart Center Bad Krozingen, Bad Krozingen, Germany

REFERENCES:
- [Result] Hochholzer W, Trenk D, Bestehorn HP, Fischer B, Valina CM, Ferenc M, Gick M, Caputo A, Buttner HJ, Neumann FJ. Impact of the degree of peri-interventional platelet inhibition after loading with clopidogrel on early clinical outcome of elective coronary stent placement. J Am Coll Cardiol. 2006 Nov 7;48(9):1742-50. doi: 10.1016/j.jacc.2006.06.065. Epub 2006 Oct 17. PMID 17084243
- [Derived] Tsimikas S, Kille A, Kaier K, Nuhrenberg T, Franke K, Valina CM, Yang X, Leibundgut G, Neumann FJ, Westermann D, Hochholzer W. Oxidized Phospholipids on ApoB-100, Platelet Activation and Reactivity, and Long-Term Cardiovascular Outcomes. Arterioscler Thromb Vasc Biol. 2025 Oct;45(10):1935-1944. doi: 10.1161/ATVBAHA.125.322347. Epub 2025 Aug 14. PMID 40808656
- [Derived] Valina CM, Merz S, Loffelhardt N, Amann M, Ferenc M, Stratz C, Neumann FJ, Hochholzer W. Risk of discontinuation of clopidogrel after 1 month following bare-metal stents: a propensity-score adjusted comparison with continued administration of clopidogrel after drug-eluting stents. J Thromb Thrombolysis. 2018 Apr;45(3):432-439. doi: 10.1007/s11239-018-1613-6. PMID 29349545
- [Derived] Hochholzer W, Valina CM, Stratz C, Amann M, Schlittenhardt D, Buttner HJ, Trenk D, Neumann FJ. High-sensitivity cardiac troponin for risk prediction in patients with and without coronary heart disease. Int J Cardiol. 2014 Sep 20;176(2):444-9. doi: 10.1016/j.ijcard.2014.07.094. Epub 2014 Aug 4. PMID 25127973
- [Derived] Trenk D, Hochholzer W, Fromm MF, Zolk O, Valina CM, Stratz C, Neumann FJ. Paraoxonase-1 Q192R polymorphism and antiplatelet effects of clopidogrel in patients undergoing elective coronary stent placement. Circ Cardiovasc Genet. 2011 Aug 1;4(4):429-36. doi: 10.1161/CIRCGENETICS.111.960112. Epub 2011 Jun 17. PMID 21685174
- [Derived] Hochholzer W, Trenk D, Fromm MF, Valina CM, Stratz C, Bestehorn HP, Buttner HJ, Neumann FJ. Impact of cytochrome P450 2C19 loss-of-function polymorphism and of major demographic characteristics on residual platelet function after loading and maintenance treatment with clopidogrel in patients undergoing elective coronary stent placement. J Am Coll Cardiol. 2010 Jun 1;55(22):2427-34. doi: 10.1016/j.jacc.2010.02.031. PMID 20510210
- [Derived] Trenk D, Hochholzer W, Fromm MF, Chialda LE, Pahl A, Valina CM, Stratz C, Schmiebusch P, Bestehorn HP, Buttner HJ, Neumann FJ. Cytochrome P450 2C19 681G>A polymorphism and high on-clopidogrel platelet reactivity associated with adverse 1-year clinical outcome of elective percutaneous coronary intervention with drug-eluting or bare-metal stents. J Am Coll Cardiol. 2008 May 20;51(20):1925-34. doi: 10.1016/j.jacc.2007.12.056. PMID 18482659